CLINICAL TRIAL: NCT01282086
Title: Evaluation of VIMA With Sevorane in Adult Patients Required General Anesthesia for Surgery in Terms of Quality of Anesthesia and Its Influence on Cardiovascular System in Common Clinical Practice (SEVOPROTECTION)
Brief Title: Evaluation of Volatile Induction and Maintenance Anesthesia (VIMA) With Sevorane in Adult Patients Requiring General Anesthesia for Surgery in Terms of Quality of Anesthesia and Its Influence on the Cardiovascular System in Common Clinical Practice
Acronym: SEVOPROTECTION
Status: Completed | Type: Observational
Sponsor: Abbott (Ukraine) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-637
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Anesthesia, General
Keywords: Sevorane; Sevoflurane; General anesthesia; Inhalation anesthesia; General surgery

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adults requiring anesthesia for surgery: Adult patients requiring general anesthesia for surgery

SUMMARY:
The main objective of this post-marketing observational study (PMOS) is to collect data of using general anesthesia in patients undergoing any surgery to create local recommendations. These data will be based on the evaluation of volatile induction and maintenance anesthesia (VIMA) with Sevorane® (sevoflurane) in adult patients requiring general anesthesia for surgery in terms of quality of anesthesia and its influence on the cardiovascular system in common clinical practice in Ukraine.

DETAILED DESCRIPTION:
This PMOS will be conducted in a prospective, multi-centre format. It is a non-interventional, observational study in which Sevorane is prescribed for adult patients undergoing general surgery for induction and maintenance of anesthesia in the usual manner in accordance with the terms of the local marketing authorization. Sevorane is used for induction and maintenance anesthesia by the choice of anesthesiologist. No additional procedures (other than standard of care) shall be applied to the patients. Each patient will be observed from the starting of anesthesia till the anesthesia end. Markers of myocardial ischemia will be detected up to the first 24 hours after anesthesia (if available). Additionally the correlation between the experience and training background of anesthesiologists and patient related outcomes of general anesthesia with sevoflurane as a single anesthetic will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing general anesthesia for planned or urgent surgery for whom Sevorane is used for induction and maintenance anesthesia by the choice of anesthesiologist

Exclusion Criteria:

* Known sensitivity to sevoflurane or other anesthetic containing halogen
* Known or suspected genetic susceptibility to malignant hyperthermia
* Receiving regional anesthetic techniques
* Receiving intravenous anesthesia
* A history of unexplained moderate/severe hepatic dysfunction with jaundice, fever, and/or eosinophilia in association with halogenated anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned or urgent surgery
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Magdik, MD, PhD, MBA, Study Director — Abbott Laboratories S.A., Ukraine
Locations (10):
- Ukraine (10):
  - Site Ref # / Investigator 49151, Dnipropetrovsk
  - Site Ref # / Investigator 49142, Kharkiv
  - Site Ref # / Investigator 52986, Kyiv
  - Site Ref # / Investigator 44445, Kyiv
  - Site Ref # / Investigator 49144, Kyiv
  - Site Ref # / Investigator 49145, Kyiv
  - Site Ref # / Investigator 49146, Lviv
  - Site Ref # / Investigator 49154, Mykolaiv
  - Site Ref # / Investigator 49148, Odesa
  - Site Ref # / Investigator 49152, Zaporizhia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults Requiring Anesthesia for Surgery
Started | 1365
Completed | 1365
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1365
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 894
  Male | 471

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Consciousness of Patients Administered Anesthesia
Description: Loss of consciousness was measured from the time the anesthetic was administered until loss of consciousness (loss of eyelash reflex) occurred.
Time Frame: Up to 16 minutes
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1343
minutes | 3.0 (1.8)

2. Primary Outcome: Time to Awakening of Patients
Description: Measured from the time anesthesia administration was stopped until the patient responded to a verbal command.
Time Frame: Every minute after anesthesia was stopped until the patient responded to a verbal command
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1359
minutes | 16.3 (38.7)

3. Primary Outcome: Time to Extubation of Patients
Description: Time to extubation was measured from the time anesthesia administration was stopped until tracheal extubation occurred.
Time Frame: Every minute after anesthesia was stopped until extubation occurred
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1359
minutes | 99.2 (481.8)

4. Primary Outcome: Anesthesiologists' Satisfaction With Using Sevorane for Induction and Maintenance Anesthesia
Description: The anesthesiologist's overall satisfaction with the inhalation anesthesia with Sevorane for each patient was assessed by means of a numerical rating scale ranging from 0 (dissatisfied) to 10 (very satisfied).
Time Frame: Day 1
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1365
units on a scale | 8.6 (1.4)

5. Primary Outcome: Patients' Overall Impression of the Anesthesia With Sevorane
Description: After awakening from anesthesia, patients were surveyed regarding their overall impression of anesthesia with Sevorane. Patients selected one of the following answers: excellent, positive, indifferent, or other.
Time Frame: Day 1
Population: All participants with available data were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1354
participants
  Excellent | 527
  Positive | 767
  Indifferent | 56
  Other | 4

6. Secondary Outcome: Systolic Blood Pressure
Description: The systolic blood pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the operation concluded.
Time Frame: Before starting anesthesia to one hour after the operation
Population: All participants with available data were included in the analysis. n= the number of participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1363
mm Hg
  Before anesthesia (n=1363) | 135.4 (17.9)
  Induction anesthesia (after intubation) (n=1362) | 116.6 (19.0)
  After surgical incision (n=1362) | 115.0 (16.7)
  After extubation (n=1360) | 123.8 (15.8)
  One hour after operation (n=1339) | 122.3 (14.5)

7. Secondary Outcome: Diastolic Blood Pressure
Description: The diastolic blood pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the operation concluded.
Time Frame: Before starting anesthesia to one hour after the operation
Population: All participants with available data were included in the analysis. n=the number of participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1364
mm Hg
  Before anesthesia (n=1364) | 83.1 (12.2)
  Induction anesthesia (after intubation) (n=1363) | 72.8 (13.5)
  After surgical incision (n=1363) | 71.6 (12.7)
  After extubation (n=1361) | 76.0 (12.2)
  One hour after operation (n=1340) | 75.1 (11.2)

8. Secondary Outcome: Mean Arterial Pressure
Description: The mean arterial pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the operation concluded.
Time Frame: Before starting anesthesia to one hour after the operation
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1341
mm Hg
  Before anesthesia (n=1341) | 101.9 (16.4)
  Induction anesthesia (after intubation) (n=1340) | 88.2 (16.4)
  After surgical incision (n=1340) | 86.8 (14.2)
  After extubation (n=1336) | 94.1 (33.5)
  One hour after operation (n=1316) | 91.7 (13.3)

9. Secondary Outcome: Heart Rate
Description: The heart rate of each patient was recorded at different time points from just before the start of anesthesia to one hour after the operation concluded.
Time Frame: Before starting anesthesia to one hour after the operation
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1363
beats per minute
  Before anesthesia (n=1363) | 83.2 (14.6)
  Induction anesthesia (after intubation) (n=1363) | 79.8 (15.4)
  After surgical incision (n=1363) | 77.4 (13.9)
  After extubation (n=1353) | 81.2 (13.2)
  One hour after operation (n=1336) | 77.5 (11.1)

10. Secondary Outcome: Presence of Deviations in Electrocardiogram Assessments During Anesthesia
Description: Electrocardiogram (ECG) assessments performed during induction of the anesthesia and maintenance were analyzed with respect to the presence of the following deviations: blockades (problems with heart electrical activity), extrasystoles (extra abnormal heart beats), arrhythmia (abnormal heart rate or rhythm), and myocardial ischemia (decreased blood flow to the heart).
Time Frame: During induction and maintenance of anesthesia on Day 1
Population: All participants with valid data were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1347
participants
  Blockades (induction) | 1
  Blockades (maintenance) | 6
  Extrasystoles (induction) | 3
  Extrasystoles (maintenance) | 20
  Arrhythmia (induction) | 5
  Arrhythmia (maintenance) | 15
  Myocardial ischemia (induction) | 0
  Myocardial ischemia (maintenance) | 8

11. Secondary Outcome: Cardiac Troponin (Troponin T) (if Available)
Description: Troponin T values measured within 24 hours of anesthesia were to be collected when available. No data were reported for this outcome measure during the study.
Time Frame: Within 24 hours after anesthesia
Population: No data were available for the cardiac troponin outcome measure.
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 0

12. Secondary Outcome: Creatine Kinase Myocardial Isoenzyme (if Available)
Description: Creatine kinase myocardial isoenzyme (CK-MB) values measured within 24 hours of anesthesia were to be collected when available.
Time Frame: Within 24 hours after anesthesia
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 47
U/L | 34.0 (12.3)

13. Secondary Outcome: Correlation Between Anesthesiologists' Clinical Experience and Hemodynamic Parameters During Anesthesia
Description: The anesthesiologists' length of clinical experience with Sevorane was collected. The influence of this experience on the changes in hemodynamic parameters during anesthesia with Sevorane was evaluated by calculating Spearman's correlation coefficient between the duration of clinical experience with Sevorane and the changes in blood pressure, mean arterial pressure, and heart rate between T0 (before anesthesia) and T1 (at the end of induction), T2 (at the end of surgical incision), T3 (at the end of extubation), T4 (1 hour after the operation), and the minimum and maximum values, respectively.
Time Frame: Before starting anesthesia to one hour after the operation
Population: as for outcome 7
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1364
Spearman's correlation coefficient
  Systolic blood pressure (T1-T0; n=1363) | -0.017
  Systolic blood pressure (T2-T0; n=1363) | -0.072
  Systolic blood pressure (T3-T0; n=1361) | -0.111
  Systolic blood pressure (T4-T0; n=1340) | -0.165
  Systolic blood pressure (Minimum-T0; n=1364) | -0.168
  Systolic blood pressure (Maximum-T0; n=1364) | -0.078
  Diastolic blood pressure (T1-T0; n=1363) | -0.054
  Diastolic blood pressure (T2-T0; n=1363) | -0.103
  Diastolic blood pressure (T3-T0; n=1361) | -0.031
  Diastolic blood pressure (T4-T0; n=1340) | -0.010
  Diastolic blood pressure (Minimum-T0; n=1364) | -0.181
  Diastolic blood pressure (Maximum-T0; n=1364) | -0.071
  Mean arterial blood pressure (T1-T0; n=1340) | -0.038
  Mean arterial blood pressure (T2-T0; n=1340) | -0.100
  Mean arterial blood pressure (T3-T0; n=1336) | -0.062
  Mean arterial blood pressure (T4-T0; n=1341) | -0.111
  Mean arterial blood pressure (Minimum-T0; n=1341) | -0.180
  Mean arterial blood pressure (Maximum-T0; n=1340) | -0.083
  Heart rate (T1-T0; n=1363) | -0.214
  Heart rate (T2-T0; n=1363) | -0.165
  Heart rate (T3-T0; n=1353) | -0.215
  Heart rate (T4-T0; n=1336) | -0.152
  Heart rate (Minimum-T0; n=1362) | -0.194
  Heart rate (Maximum-T0; n=1358) | -0.222

14. Secondary Outcome: Correlation Between Anesthesiologists' Clinical Experience and Time to Extubation and Awakening
Description: Anesthesiologists' length of clinical experience with general anesthesia and modern inhalation agents was collected. The influence of this clinical experience on anesthesia parameters was evaluated by calculating Spearman's correlation coefficient between the duration of clinical experience (exp) with inhalation (inh) anesthesia and Sevorane on the time to extubation and the time to awakening, respectively.
Time Frame: Every minute after anesthesia was stopped until the patient was extubated and until the patient responded to a verbal command.
Population: All participants with available data at each time point were included in the analysis.
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1359
Spearman's correlation coefficient
  Exp w/ inh anesthesia (time to extubation) | 0.019
  Exp w/ inh anesthesia (time to awakening) | -0.142
  Exp w/ Sevorane (time to extubation) | 0.016
  Exp w/ Sevorane (time to awakening) | 0.211

ADVERSE EVENTS:
Time Frame: Physicians were to report all adverse events occurring during the induction phase, maintenance phase, and recovery phase of surgery.
Arm/Group | Adults Requiring Anesthesia for Surgery
Serious Adverse Events (participants affected / at risk) | 2/1365
Other Adverse Events (participants affected / at risk) | 7/1365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults Requiring Anesthesia for Surgery (N=1365)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Operative Hemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults Requiring Anesthesia for Surgery (N=1365)
Unwanted Awareness During Anesthesia (Injury, poisoning and procedural complications) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cognitive Disorders (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hyperthermia (General disorders) | 1
Psychomotor Hyperactivity (Psychiatric disorders) | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The data on troponin T values were not collected in the study and CK-MB was detected in a small number of patients, therefore no conclusions can be made regarding the influence of VIMA with Sevorane on myocardial ischemia markers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.